CLINICAL TRIAL: NCT05382780
Title: Effect of Breather Trainer Versus Pulmonary Rehabilitation on Cardiopulmonary Efficiency in Patients With COPD Post COVID-19
Brief Title: Breather Trainer Versus Pulmonary Rehabilitation on Cardiopulmonary Efficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Eman Rashad Ali Elsayed, Principal investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Eman_Rashad_PhD_2022
Record Dates: First submitted 2022-04-24; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; COPD
MeSH Terms: conditions — COVID-19; Pulmonary Disease, Chronic Obstructive | interventions — Contraceptive Devices, Female

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The breather respiratory muscle trainer group (Experimental): 40 patients (20 males and 20 females) will receive The breather respiratory muscle trainer for 30 minutes and mild interval aerobic training and respiratory training on treadmill 3 times / week for 12 weeks.
  Interventions: Other: The breather respiratory muscle trainer; Other: interval aerobic training and respiratory training
- Diaphragmatic and localized breathing exercises group (Experimental): 40 patients (20 males and 20 females) will receive diaphragmatic and localized breathing exercises ( especially Middle & Lower segments) and mild intensity interval aerobic training and respiratory training on treadmill 3 times / week for 12 weeks,
  Interventions: Other: Diaphragmatic and localized breathing exercises; Other: interval aerobic training and respiratory training

INTERVENTIONS:
Other: The breather respiratory muscle trainer — The breather respiratory muscle training device is a high quality and effective trainer designed to specifically train the inspiratory and expiratory muscles in one same breathing action. The device allows for adjustable levels of resistance using easy-to-read dials, which allows you to adjust the device to the settings you require. The inhale settings allow for adjustment 1-6 with 1 being the easiest and 6 being the hardest, while the exhale settings allow for adjustment 1-5, where 1 in the easiest and 5 the hardest.
  Arms: The breather respiratory muscle trainer group
Other: Diaphragmatic and localized breathing exercises — A. Diaphragmatic breathing exercises:
  Exercise will be performed as prescribed in the clinical guidelines for 5-10 minutes about 3-4 times per day.
  B. Localized Breathing:
  Exercise will be performed as prescribed in the clinical guidelines for 5-10 minutes about 3-4 times per day.
  C. Mild Interval training exercise
  Arms: Diaphragmatic and localized breathing exercises group
Other: interval aerobic training and respiratory training — mild intensity interval aerobic training and respiratory training on treadmill

SUMMARY:
The purpose of the study is to determine the difference between The Breather respiratory muscle trainer and pulmonary rehabilitation in patients with COPD post COVID-19.

DETAILED DESCRIPTION:
The main concern in post COVID-19 patients is the involvement of respiratory system and cardiovascular system which may result in dyspnea, low blood oxygen saturation, and decrease cardiopulmonary efficiency.

In cases of post COVID-19 patients with COPD their state is deconditioned and more critical than normal to be either in the zone of progression or regression or stability as the studies showed that handling of these cases during (3-6 months post-COVID) will prevent these symptoms from becoming permanent.

ELIGIBILITY:
Inclusion Criteria:

1. SPO2 ≥ 93%
2. Their age ranges from 30-40 years old.
3. COPD patients GOLD1 (Mild FEV1≥80% predicted) and GOLD2 (Moderate 50% ≤FEV1<80%predicted) (Manian, 2019)
4. patients diagnosed as post COVID-19 Pneumonia between 3 and 6 Months ago with CT scan and PCR testing.
5. Their body mass index (BMI) ranged from 20 to 29.9kg/m2.
6. Stable medical cases with dyspnea

Exclusion Criteria:

Patients who will meet one of the following criteria will be excluded from the study:

1. patients with cardiac problems e.g. atrial fibrillation, left bundle-branch block, heart failure.
2. Sever cases of COPD (FEV1/FVC< 50%)
3. Mitral or aortic valvular disease, pericardial effusion.
4. Recent myocardial infarction.

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of change in Physical Fitness Index (PFI) | at baseline and 3 months of intervention
  To assess the change in Physical Fitness Index (PFI) By using Modified Harvard Step Test (HST): The test will be done on a step height of 33 cm height. PFI was calculated by using following formula
Assessment of change in Rate Pressure Product | at baseline and 3 months of intervention
  To assess the change in Rate Pressure Product. First, the baseline heart rate (HR), systolic blood pressure (SBP) and diastolic blood pressure (DBP) will be recorded, by an aneroid sphygmomanometer. HR will be constantly displayed on pulse oximetry.
  The rate-pressure product (RPP) = HR X SBP
Assessment of change in Forced vital capacity | at baseline and 3 months of intervention
  To assess the change in Forced vital capacity (FVC) by spirometry. The unit of measure is liters.
Assessment of change in Forced expiratory volume in the first one second | at baseline and 3 months of intervention
  To assess the change in Forced expiratory volume in the first one second (FEV1) by spirometry. The unit of measure is liters.
Assessment of change in Ratio of forced expiratory volume in the first one second to the forced vital capacity of lungs | at baseline and 3 months of intervention
  To assess the change in the ratio of forced expiratory volume in the first one second to the forced vital capacity of lungs (FEV1/FVC) by spirometry. The unit of measure is the ratio.
Assessment of change in Maximum voluntry ventilation | at baseline and 3 months of intervention
  To assess the change in the maximum voluntary ventilation (MVV) by spirometry. The unit of measure is the liters/ minute.
Assessment of change in Forced vital capacity expressed as percentage of the predicted FVC | at baseline and 3 months of intervention
  To assess the change in the Forced vital capacity expressed as a percentage of the predicted FVC (FVC%) by spirometry. The unit of measure is the liters.
Assessment of change in Forced expiratory volume in the first one second expressed as percentage of the predicted FEV1 | at baseline and 3 months of intervention
  To assess the change in the Forced expiratory volume in the first one second expressed as a percentage of the predicted FEV1 (FEV1%) by spirometry. The unit of measure is the liters.

SECONDARY OUTCOMES:
Assessment of change in Oxygen saturation | at baseline and 3 months of intervention
  To assess the change in the Oxygen saturation using pulse oximeter device.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Rashad, Assistant lecturer, Principal Investigator — Horus University in Egypt
Locations (1):
- Outpatient clinic, Faculty of Physical Therapy, Horus University, Egypt, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided